CLINICAL TRIAL: NCT04615598
Title: Evaluation of the Effects of Action Observation Training on Tongue Strength in Brain-damaged Patients: a Non-randomized Controlled Trial
Brief Title: Assessment of the Effects of Mental Practice on Tongue Strength in Brain-damaged Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: uammadrid91
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Movement, Involuntary
Keywords: Action observation
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action observation group (Experimental)
  Interventions: Behavioral: Action observation
- Placebo group (Placebo Comparator)
  Interventions: Behavioral: Placebo group

INTERVENTIONS:
Behavioral: Action observation — The idea is to show some videos with the aim of improving patients' tongue strength.
  Arms: Action observation group
Behavioral: Placebo group — The idea is to show some videos of vegetation with the aim of having an intervention time but ineffective.
  Arms: Placebo group

SUMMARY:
The main objective is to evaluate the effects of action-observation training on tongue strength in brain-damaged patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Date of injury : 6 months onwards
* Medical diagnosis: brain damage or head trauma
* Clinical diagnosis of dysphagia by videofluoroscopy or V-CAM and expert opinion.

Exclusion Criteria:

* Not understanding verbal or auditory/visual commands through the Boston Test
* Present behavioural alterations
* Presence of seizures
* Presence of tracheotomy
* Impulsivity
* Attention Problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Lingual strength | Change in immediately at the end of the intervention and also, changes between the end and three months
  The IOPI instrument has a mechanical sensor that evaluates the force.

SECONDARY OUTCOMES:
Cervical Range of motion | Change in immediately at the end of the intervention and also, changes between the end and three months
  The cervical goniometer will measure the active cervical range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain